CLINICAL TRIAL: NCT03606278
Title: Evaluation of Two Strategies for Constructive Immediate Feedback in the Development of Skills for Neonatal Resuscitation: a Randomized Clinical Trial
Brief Title: Evaluation of Two Strategies for Debriefing in the Development of Skills for Neonatal Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de la Sabana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Acta 366 11-Dic-2015
Record Dates: First submitted 2018-07-13; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Asphyxia Neonatorum; Birth Injuries; Cardiopulmonary Resuscitation
Keywords: Debriefing
MeSH Terms: conditions — Asphyxia Neonatorum; Birth Injuries

STUDY DESIGN:
Intervention Model Description: The study participants were randomly assigned to the type of debriefing (oral or video), stratified by the type of health professional. For this randomization, the random function of Excel was used, sorting the participants in a random number order and assigning the first half to the oral group and the other half to the video-assisted group. For the conformation of the teams, a second randomization was performed, in which the professionals within an assigned group (oral or video-assisted) were randomized to form a resuscitation team. In this randomization, Excel's random function was also used, sorting the patients in a random number order and assigning the one that was ordered first to team 1, the second to team 2, and so on, each team had three professions: pediatrician, professional nurse, and respiratory therapist. The same team was maintained during the participation of each scenario.
Who Masked: Outcomes Assessor
Masking Description: For the performance and evaluation score of the adherence of the teams to the resuscitation protocols, a review of the literature was performed, and the modified version of the validated Neonatal Resuscitation Performance Evaluation (NRPE) tool was considered (1). Given that this instrument did not consider behavioral and leadership aspects, a checklist of individual performance and performance by profession was constructed in each of the scenarios that included cognitive/technical and behavioral aspects. This checklist was applied by a reviewer blinded to the assignment of the type of debriefing by reviewing the video of the participation of the groups in the scenarios.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured debriefing assisted by video (Experimental): In the structured debriefing assisted by video, the process was based on the immediate review of the video, stopping and rewinding the recording as required.
  Interventions: Other: Structured debriefing assisted by video
- Structured oral debriefing (Active Comparator): In the structured oral debriefing, the process was based by the mental search of their memories of what occurred.
  Interventions: Other: Structured oral debriefing

INTERVENTIONS:
Other: Structured debriefing assisted by video — In the structured debriefing assisted by video, the process was based on the immediate review of the video, stopping and rewinding the recording as required. The debriefing session was conducted in the debriefing room of the simulation laboratory with an assigned time of 15 minutes. Each session was developed in three phases. The first phase, descriptive, in which each participant was encouraged to recount what they had lived and experienced, clarifying how the events unfolded, verifying the appropriate decisions and the errors committed in the scenario and the ways they could have solved them and corrected them. The second phase, analytical, the participant reflected on what occurred in the scenario, commenting on how their feelings were involved in the development of the case. The third phase, application or transference, in which the group was encouraged to draw conclusions from what had occurred, realizing an application of this experience in a real-life.
  Arms: Structured debriefing assisted by video
Other: Structured oral debriefing — In the structured oral debriefing, the process was based by the mental search of their memories of what occurred. The debriefing session was conducted in the debriefing room of the simulation laboratory with an assigned time of 15 minutes. Each session was developed in three phases. The first phase, descriptive, in which each participant was encouraged to recount what they had lived and experienced, clarifying how the events unfolded, verifying the appropriate decisions and the errors committed in the scenario and the ways they could have solved them and corrected them. The second phase, analytical, the participant reflected on what occurred in the scenario, commenting on how their feelings were involved in the development of the case. The third phase, application or transference, in which the group was encouraged to draw conclusions from what had occurred, realizing an application of this experience in a real-life.
  Arms: Structured oral debriefing

SUMMARY:
Introduction: Training of health professionals in neonatal resuscitation reduces risks and adverse events during this intervention. Simulation-based education with constructive immediate feedback (debriefing) is an effective teaching method for personnel in charge of neonatal resuscitation.

Objective: To evaluate two debriefing strategies for the development of neonatal resuscitation skills in professionals specialized in critical newborn care.

Materials and Methods: A simple blind randomized clinical trial was conducted. Twenty-four professionals (pediatricians, nurses, and respiratory therapists) were randomly assigned for two interventions; one group received oral debriefing and the other oral debriefing assisted by video. Three standardized clinical scenarios that were recorded on video were executed. A checklist was applied for the evaluation, administered by a reviewer blinded to the assignment of the type of debriefing.

Null hypothesis: The improved in the skills of neonatal resuscitation is the same for both strategies of debriefing.

Alternative hypothesis: The improved in the skills of neonatal resuscitation is different for both strategies of debriefing

ELIGIBILITY:
Inclusion Criteria:

* The specialized health professionals (Professional nurses, respiratory therapists, and pediatricians) in charge of newborn care that working in the Neonatal Unit areas, maternity wards, surgery rooms responsible for the care of caesarean sections, and those of pediatric emergencies of University Hospital of La Sabana

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Compliance percentage of the activities | The checklist was applied by a reviewer blinded to the assignment of the type of debriefing by reviewing the video, on average 1 week after of the participation of the groups in the scenarios.
  For the performance and evaluation score of the adherence of the teams to the resuscitation protocols, a review of the literature was performed for constructed a checklist that included cognitive/technical and behavioral aspects of individual performance and performance by profession in each of the scenarios. Each item of the tool was assigned a score of 1 if the evaluated activity was correctly performed, 0 if it was not performed correctly, and N/A if it did not apply for the scenario and/or for the profession. A compliance percentage (range 0% to 100%) of the activities evaluated by participant in the tool was obtained, summed the points obtained onto the possible total score. The higher percentage indicate better outcome.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Sawyer T, Sierocka-Castaneda A, Chan D, Berg B, Lustik M, Thompson M. Deliberate practice using simulation improves neonatal resuscitation performance. Simul Healthc. 2011 Dec;6(6):327-36. doi: 10.1097/SIH.0b013e31822b1307. PMID 21937960
- [Derived] Gamboa OA, Agudelo SI, Maldonado MJ, Leguizamon DC, Cala SM. Evaluation of two strategies for debriefing simulation in the development of skills for neonatal resuscitation: a randomized clinical trial. BMC Res Notes. 2018 Oct 17;11(1):739. doi: 10.1186/s13104-018-3831-6. PMID 30333050